CLINICAL TRIAL: NCT00665158
Title: Prevention and Reduction of Obesity Through Active Living
Acronym: PROACTIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Bob Ross, Professor, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ross2006
Record Dates: First submitted 2008-04-21; First posted 2008-04-23 (Estimated); Last update posted 2011-10-31 (Estimated); Status verified 2008-10

CONDITIONS: Obesity
Keywords: Abdominal obesity, exercise, behaviour modification
MeSH Terms: conditions — Obesity; Obesity, Abdominal; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- UC (Active Comparator): Usual Care Group
  Interventions: Behavioral: UC (Usual Care Group)
- BI (Active Comparator): Behavioural Intervention Group
  Interventions: Behavioral: BI (Behavioral Intervention Group)

INTERVENTIONS:
Behavioral: UC (Usual Care Group) — Usual Care Group - Treatment Implementation by Primary Care Physician
  Arms: UC
Behavioral: BI (Behavioral Intervention Group) — Behavioral Intervention Group - Treatment Implementation by Health Educator
  Arms: BI

SUMMARY:
We will perform a randomized, controlled trial, the primary aim of which is to assess the effectiveness of a behavioral-based physical activity program in the prevention and treatment of obesity and related co-morbid conditions in a primary care setting. We hypothesize that the prevention and/or reduction of obesity and related co-morbidities in patients randomized to an individualized education and behavior counseling group will be greater by comparison to those randomized to a group that receives standard care alone.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 25 and 65 years of age.
* Sedentary lifestyle (planned physical activity for the purpose of health one day per week or less).
* Abdominally obese (waist circumference greater than 88 and 102 cm for women and men respectively).
* Weight stable (± 2 kg) for 6 months prior to the beginning of the study.
* BMI between 25 and 34.9 kg/m2 (Because a lifestyle-based intervention alone for obesity reduction is ideal for persons with a BMI greater less than 35, and, that 94% of overweight and obese Canadian adults have a BMI between 25 and 34.9 kg/m2, subjects with a BMI 35 or greater will be excluded).

Exclusion Criteria:

* Physical impairment which would make the intervention very difficult, or unsafe according to the patient's physician including history of myocardial infarction, stroke, coronary bypass surgery or angioplasty in the last 6 months; peripheral artery disease, unstable angina or ischemia, uncontrolled or insulin dependent diabetes mellitus.
* Alcohol consumption > 21 drinks per week.
* Plans to move from the area.
* Participating in another research study.
* Clinically judged to be unsuitable for participation or adherence
* Inability or unwillingness to provide informed consent.
* For women, planned pregnancy in the next 3 years.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2003-09; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Waist Circumference | 2 Years

SECONDARY OUTCOMES:
Metabolic Syndrome | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Robert Ross, Principal Investigator — Queen's University
Locations (1):
- Queen's University : Physical Education Center, Kingston, Ontario, Canada

REFERENCES:
- [Derived] Ross R, Lam M, Blair SN, Church TS, Godwin M, Hotz SB, Johnson A, Katzmarzyk PT, Levesque L, MacDonald S. Trial of prevention and reduction of obesity through active living in clinical settings: a randomized controlled trial. Arch Intern Med. 2012 Mar 12;172(5):414-24. doi: 10.1001/archinternmed.2011.1972. Epub 2012 Feb 27. PMID 22371872